CLINICAL TRIAL: NCT00694369
Title: A Phase III Randomized, Double-Blind, Placebo- and Active-Comparator-Controlled Multiple-Dose Clinical Trial to Study the Efficacy and Safety of MK0663/Etoricoxib 90 and 120 mg, Ibuprofen 600 mg, and Acetaminophen 600 mg/Codeine 60 mg in the Treatment of Patients With Postoperative Dental Pain
Brief Title: A Study to Asses the Effect of MK0663 in the Treatment of Patients With Postoperative Dental Pain (0663-092)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-092; MK0663-092; 2008_506
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Results first posted 2010-01-29 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Postoperative Dental Pain
Keywords: Postoperative Dental Pain
MeSH Terms: interventions — Codeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): etoricoxib 90 mg
  Interventions: Drug: Comparator: etoricoxib
- 2 (Experimental): etoricoxib 120 mg
  Interventions: Drug: Comparator: etoricoxib
- 3 (Active Comparator): ibuprofen 2400 mg
  Interventions: Drug: Comparator: ibuprofen
- 4 (Active Comparator): acetaminophen 2400 mg/codeine 240 mg
  Interventions: Drug: Comparator: acetaminophen + codeine
- 5 (Placebo Comparator): Matching Placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: Comparator: etoricoxib — etoricoxib 90 mg; 120 mg (once daily) over three days.
  Arms: 1; 2
Drug: Comparator: ibuprofen — ibuprofen 2400 mg (600 mg Q6h) over three Days
  Arms: 3
Drug: Comparator: acetaminophen + codeine — acetaminophen 2400 mg/codeine 240 mg (600/60 mg Q6h) over three Days
  Arms: 4
Drug: Comparator: placebo — matching placebo over three Days
  Arms: 5

SUMMARY:
The purpose of this study is to compare the pain relieving effect of different doses of MK0663 with placebo and other pain relievers/analgesics in patients with postoperative dental pain. Pain intensity and relief will be measured by the total pain relief score (TOPAR) and patient evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be scheduled to have 2 or more third molars removed, at least 1 of which is partially embedded in bone and is impacted in the lower jaw
* Patients must be experiencing moderate to severe pain following the dental procedure

Exclusion Criteria:

* Previous molar extraction within the past 45 days
* Personal or family history of an inherited bleeding disorder
* Uncontrolled high blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Brown JD, Daniels SE, Bandy DP, Ko AT, Gammaitoni A, Mehta A, Boice JA, Losada MC, Peloso PM. Evaluation of multiday analgesia with etoricoxib in a double-blind, randomized controlled trial using the postoperative third-molar extraction dental pain model. Clin J Pain. 2013 Jun;29(6):492-8. doi: 10.1097/AJP.0b013e318260c144. PMID 23247002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Conducted at 3 investigational sites in the US. Patients were recruited from the sites patient pool and through advertising. A total of 588 patients were randomized. First Patient Entered 27-June-2008; First Patient In (randomized) on 03-July- 2008; Last Patient Last Visit 08-Jan-09
Pre-assignment Details: Patients who met entry criteria and were experiencing moderate-to-severe pain after removal of at least 2
  third molars (at least 1 being partially or completely impacted and of mandibular origin) were allocated to
  the study. Wash-out period for exclusionary medication was specified in the protocol. Randomization was
  stratified by baseline pain.
Groups:
- Placebo: Placebo orally once daily
- Etoricoxib 90 mg: Etoricoxib 90 mg orally once daily
- Etoricoxib 120 mg: Etoricoxib 120 mg orally once daily
- Ibuprofen 2400 mg: Ibuprofen 2400 mg (600 mg every 6 hours (Q6h)) orally
- Acetaminophen 2400 mg/Codeine 240 mg: Acetaminophen 2400 mg/Codeine 240 mg (600/60 mg Q6h) orally
Period: Overall Study
Arm/Group | Placebo | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 2400 mg | Acetaminophen 2400 mg/Codeine 240 mg
Started | 46 | 191 | 97 | 192 | 62
Completed | 45 | 188 | 95 | 189 | 56
Not Completed | 1 | 3 | 2 | 3 | 6
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 2400 mg | Acetaminophen 2400 mg/Codeine 240 mg | Total
Number analyzed (Participants) | 46 | 191 | 97 | 192 | 62 | 588
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.0 (3.0) | 21.8 (3.6) | 21.8 (3.5) | 21.6 (3.8) | 20.5 (2.8) | 21.5 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 113 | 50 | 115 | 37 | 340
  Male | 21 | 78 | 47 | 77 | 25 | 248
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 52 | 25 | 50 | 17 | 155
  Not Hispanic or Latino | 35 | 139 | 72 | 142 | 44 | 432
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 1 | 1 | 5
  Asian | 0 | 6 | 4 | 9 | 0 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 1 | 1 | 4
  Black or African American | 2 | 4 | 1 | 7 | 3 | 17
  White | 43 | 174 | 86 | 173 | 56 | 532
  More than one race | 1 | 5 | 3 | 1 | 1 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Baseline Pain Intensity [Number; unit: Participants] — The level of pain at baseline (before dosing) is indicated by the patient on the patient diary by placing a check mark next to the appropriate response to the following question (My starting pain is: None, Slight, Moderate, Severe). Patients who indicated moderate to severe pain at baseline were eligible to be
  randomized into the study.
  Participants
    Moderate | 21 | 98 | 49 | 106 | 30 | 304
    Severe | 25 | 93 | 48 | 86 | 32 | 284
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 71.21 (16.33) | 72.53 (16.68) | 71.02 (15.96) | 72.24 (16.81) | 69.43 (13.99) | 71.76 (16.29)
Duration of Surgery [Mean (Standard Deviation); unit: Hours] | 0.14 (0.06) | 0.13 (0.06) | 0.15 (0.08) | 0.14 (0.06) | 0.13 (0.06) | 0.14 (0.06)
Height [Mean (Standard Deviation); unit: Centimeters] | 171.03 (8.91) | 168.39 (9.95) | 167.92 (10.07) | 168.50 (9.05) | 168.38 (9.86) | 168.56 (9.59)
Mean Impaction Score [Mean (Standard Deviation); unit: Units on a Scale] — Impaction Score (Soft Tissue =1, Partial Embedded= 2,
  Embedded = 3)
  Units on a Scale | 2.41 (0.51) | 2.44 (0.50) | 2.40 (0.52) | 2.50 (0.48) | 2.40 (0.51) | 2.45 (0.50)
Number of Hours from End of Surgery to Dosing [Mean (Standard Deviation); unit: Hours] | 3.06 (0.79) | 2.94 (0.77) | 2.84 (0.75) | 3.01 (0.84) | 2.97 (0.78) | 2.96 (0.79)
Number of Teeth Removed [Mean (Standard Deviation); unit: Teeth] | 2.04 (0.29) | 2.06 (0.27) | 2.10 (0.39) | 2.02 (0.12) | 2.03 (0.18) | 2.05 (0.26)

OUTCOME MEASURES:

1. Primary Outcome: Total Pain Relief Score Over the First 6 Hours Post the Initial Day 1 Dose of the Study Medication (TOPAR6)
Description: TOPAR6 was calculated by multiplying the pain relief (PR) score (0- to 4-point Likert scale, with 0=None, and 4=Complete for pain relief) at each time point by the duration (in hours) since the preceding time point, and summing these weighted values up to 6 hours post the initial Day 1 dose. The range of TOPAR6 score is 0 to 24.
Time Frame: Over the first 6 hours post the initial Day 1 dose of the study medication
Population: Full Analysis Set population (all randomized patients who received at least 1 dose of study treatment and had at least 1 post-baseline PR data over the first 6 hours). Observed PR was used up to rescue. Missing data was imputed by linear interpolation at time points before rescue, by last-observation-carried-forward at time points after rescue.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 2400 mg | Acetaminophen 2400 mg/Codeine 240 mg
Number analyzed (Participants) | 46 | 191 | 97 | 192 | 62
Units on a Scale | 5.08 (0.86) | 16.10 (0.42) | 15.73 (0.59) | 15.67 (0.42) | 11.83 (0.74)
Statistical Analysis 1: Comparison: Placebo vs Etoricoxib 120 mg; Test type: Superiority or Other; p < 0.001, ANOVA — 0.05 critical level was used; Step-down manner was used (p-value for 90-mg dose comparison was reported only if the p-value for 120-mg dose comparison is significant)
Statistical Analysis 2: Comparison: Placebo vs Etoricoxib 90 mg; Test type: Superiority or Other; p < 0.001, ANOVA — 0.05 critical level was used; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Etoricoxib 120 mg vs Ibuprofen 2400 mg; Test type: Non-Inferiority or Equivalence — Non-inferiority bound (etoricoxib minus ibuprofen) is -4.45; Difference in LS Means = 0.06, 95% CI [-1.37 to 1.48] — Difference in Least squares means (LS Means) (etoricoxib minus ibuprofen)
Statistical Analysis 4: Comparison: Etoricoxib 90 mg vs Ibuprofen 2400 mg; Test type: Non-Inferiority or Equivalence — Non-inferiority bound (etoricoxib minus ibuprofen) is -4.45; Difference in LS Means = 0.43, 95% CI [-0.73 to 1.60] — Difference in LS Means (etoricoxib minus ibuprofen)
Statistical Analysis 5: Comparison: Etoricoxib 120 mg vs Acetaminophen 2400 mg/Codeine 240 mg; Test type: Non-Inferiority or Equivalence — Non-inferiority bound (etoricoxib minus cetaminophen/codeine) is -2.41; Difference in LS Means = 3.90, 95% CI [2.04 to 5.76] — Difference in LS Means (etoricoxib minus acetaminophen/codeine)
Statistical Analysis 6: Comparison: Etoricoxib 90 mg vs Acetaminophen 2400 mg/Codeine 240 mg; Test type: Non-Inferiority or Equivalence — Non-inferiority bound (etoricoxib minus acetaminophen/codeine) is -2.41; Difference in LS Means = 4.27, 95% CI [2.61 to 5.94] — Difference in LS Means (etoricoxib minus acetaminophen/codeine)
Statistical Analysis 7: Comparison: Etoricoxib 90 mg vs Etoricoxib 120 mg; Test type: Superiority or Other; Difference in LS Means = -0.38, 95% CI [-1.80 to 1.05] — Difference in LS Means (etoricoxib 120 mg minus etoricoxib 90 mg)
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 2400 mg; Test type: Superiority or Other; Difference in LS Means = 10.59, 95% CI [8.72 to 12.47] — Difference in LS Means (ibuprofen 2400 mg minus placebo)
Statistical Analysis 9: Comparison: Placebo vs Acetaminophen 2400 mg/Codeine 240 mg; Test type: Superiority or Other; Difference in LS Means = 6.75, 95% CI [4.53 to 8.97] — Difference in LS Means (acetaminophen 2400 mg/codeine 240 mg minus placebo)

2. Secondary Outcome: Patient's Global Assessment of Study Medication at 24 Hours Post the Initial Day 1 Dose of the Study Medication
Description: Patient's Global Assessment of Study Medication was on 0- to 4- point scale, with 0=Poor, and 4=Excellent for patient's rating of the study medication for pain.
Time Frame: At 24 hours post the initial Day 1 dose of the study medication
Population: Full Analysis Set population (all randomized patients who received at least 1 dose of study treatment and had at least 1 post-baseline assessment at 24 hours). Observed data was used. Forty patients were excluded from the analysis due to no measurement at 24 hours after the initial Day 1 dose.
Measure: Number; unit: Participants
Arm/Group | Placebo | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 2400 mg | Acetaminophen 2400 mg/Codeine 240 mg
Number analyzed (Participants) | 44 | 184 | 86 | 180 | 54
Participants
  Poor | 19 | 12 | 7 | 6 | 1
  Fair | 12 | 12 | 5 | 24 | 13
  Good | 5 | 43 | 20 | 42 | 15
  Very Good | 5 | 66 | 26 | 73 | 18
  Excellent | 3 | 51 | 28 | 35 | 7
Statistical Analysis 1: Comparison: Placebo vs Etoricoxib 120 mg; Test type: Superiority or Other; p < 0.001, stratified Wilcoxon rank sum test — 0.05 critical level was used; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Etoricoxib 90 mg; Test type: Superiority or Other; p < 0.001, stratified Wilcoxon rank sum test — 0.05 critical level was used; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Etoricoxib 120 mg vs Ibuprofen 2400 mg; Test type: Superiority or Other; p = 0.161, stratified Wilcoxon rank sum test — 0.05 critical level was used; Nominal p-value was provided in lieu of the 95% CI. Step-down manner was used, and the nominal p-value for 90-mg dose comparison was not reported
Statistical Analysis 4: Comparison: Etoricoxib 120 mg vs Acetaminophen 2400 mg/Codeine 240 mg; Test type: Superiority or Other; p = 0.014, stratified Wilcoxon rank sum test — 0.05 critical level was used; Nominal p-value was provided in lieu of the 95% CI. Step-down manner was used
Statistical Analysis 5: Comparison: Etoricoxib 90 mg vs Acetaminophen 2400 mg/Codeine 240 mg; Test type: Superiority or Other; p = 0.007, stratified Wilcoxon rank sum test — 0.05 critical level was used; Nominal p-value was provided in lieu of the 95% CI. Step-down manner was used

ADVERSE EVENTS:
Time Frame: Adverse experiences were collected from the Pre-surgery/Pre-treatment period through the 14 day safety follow-up period.
Arm/Group | Placebo | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 2400 mg | Acetaminophen 2400 mg/Codeine 240 mg
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/191 | 0/97 | 0/192 | 0/62
Other Adverse Events (participants affected / at risk) | 12/46 | 54/191 | 28/97 | 57/192 | 35/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | Etoricoxib 90 mg (N=191) | Etoricoxib 120 mg (N=97) | Ibuprofen 2400 mg (N=192) | Acetaminophen 2400 mg/Codeine 240 mg (N=62)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 2 | 0
Blepharospasm (Eye disorders) | 1 | 0 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 2 | 0
Visual Impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 6 | 4 | 10 | 23
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 15
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 0 | 1 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0
Alveolar osteitis (Infections and infestations) | 0 | 8 | 3 | 8 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 4 | 0 | 3 | 10
Dysgeusia (Nervous system disorders) | 0 | 2 | 3 | 0 | 0
Headache (Nervous system disorders) | 6 | 11 | 5 | 8 | 9
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 4 | 2 | 6 | 5
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Flushing (Vascular disorders) | 2 | 0 | 1 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.